CLINICAL TRIAL: NCT04045197
Title: The Effect of Relaxation-Focused Nursing Care on Stress, Cortisol and Birth Week in Threat of Preterm Birth: A Randomised Controlled Trial
Brief Title: Nursing Care in Threat of Preterm Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hülya Özberk (Other)
Collaborators: Dokuz Eylul University (Other)
Responsible Party: Sponsor-Investigator, Hülya Özberk, Research Assistant,Deparment of Obstetric-Women's Diseases Nursing,Principal Investigator, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DokuzEU12345
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Nursing Caries
Keywords: Relaxation

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Participant
Masking Description: Single Blind Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In the intervention group; informed consent forms, Relaxation Focused Nursing Care and routine nursing care in the hospital were performed. Then data collection tools were applied.
  Interventions: Behavioral: Relaxation Focused Nursing Care
- Control group (No Intervention): Women in the control group received routine nursing care in the hospital and data collection tools were applied at the same hours as the intervention group.

INTERVENTIONS:
Behavioral: Relaxation Focused Nursing Care — "Relaxation Focused Nursing Care" is composed of HypnoBirthing and Transactional Model. Hypnobirthing Philosophy is based on the laws of mind and aims to create positive thoughts and emotions. The Transactional Model defines stress as a special relationship between the person and the environment. Therefore, Relaxation Focused Nursing Care; positive language, positive environment and reducing stressors.
  Other Names: Information
  Arms: Intervention group

SUMMARY:
Relaxation-Focused Nursing Care which is formed by using these two models is composed of; positive language, positive environment and reducing stressors. Relaxation-Focused Nursing Care, which is thought to have an effect on delaying birth, consists of four stages as a two-day program.In this study, it is aimed to determine the effect of Relaxation-Focused Nursing Care on stress level, cortisol level and birth week.

DETAILED DESCRIPTION:
Preterm birth is seen in 7-12% of all pregnant women and according to estimations about 15 million infants are delivered each year. Preterm birth is an extremely important problem in terms of its effects on newborn's health, mother's health, community and economy. Preterm birth causes the newborn chronic pulmonary disease; gastrointestinal, immunologic, central nervous system, auditory and visual problems; long-term motor and cardiovascular system diseases; and cognitive, visual, behavioral disorders. While preterm birth causes the women postpartum anxiety, stress and depression; it also leads to newborn intensive care costs, long-term complex health care needs for families and community and has serious consequences for public service sector such as health insurance, education, other social support systems and economy. Some factors initiate preterm birth, whereas 70-80% of them start spontaneously, remaining 20-30% has iatrogenic origin. It is reported that there is no known and effective treatment for preterm birth. It is reported in literature that stress which is one of the risk factors of preterm birth, causes preterm birth. If stress causes threat of preterm delivery, reducing stress may delay preterm birth and the complications of preterm birth on newborn and mother's health and also its economic and social burden can be reduced. National and international studies related to the effect of coping with stress on threat of preterm birth are lacking. It is thought that preterm birth can be prevented in women with threat of preterm birth through developing mechanisms to cope with stress and reducing stressors. Since nurse provides 24-hour care for woman diagnosed with the threat of preterm birth, the nursing care may be effective in this aspect.

ELIGIBILITY:
Inclusion Criteria:

* to be diagnosed with TPB,
* to be over 18 years of age,
* to know Turkish and
* to agree to participate in the research.

Exclusion Criteria:

* diagnosis of EMR,
* multiple pregnancy,
* admission to hospital with vaginal bleeding,
* psychiatric, chronic and pregnancy-related disease developing,
* to want to quit the study at any stage after agreeing to participate in the study, and
* delivery at any stage after the data collection process has been completed after agreeing to participate in the trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — To be over 18 years of age
Enrollment: 66 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Birth weeks of Intervention and Control Groups | 20 weeks
  Comparison of birth weeks between intervention and control groups

SECONDARY OUTCOMES:
Stress level of Intervention and Control Groups | 2 days
  Comparison of stress level between intervention and control groups, physiological parameter

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Özberk, PhD, Principal Investigator — Dokuz Eylul University; Samiye Mete, PhD, Study Director — University of Kyrenia; Murat Bektaş, PhD, Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)